CLINICAL TRIAL: NCT05547893
Title: Clinical Learning Through Extended Immersion in Medical Simulation (CLEIMS)-A New Approach to Teaching Clinical Ethics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KMUHIRB-SV(II)-20200041
Record Dates: First submitted 2022-09-04; First posted 2022-09-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Educational Activities; Patient Simulation
Keywords: medical ethics education; simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): workshop discussing the clinical ethical case scenario
- Intervention group (Experimental): a simulated clinical ethical situation with simulation patients
  Interventions: Other: simulation

INTERVENTIONS:
Other: simulation — participating a simulated clinical ethical situation with simulation patients
  Arms: Intervention group

SUMMARY:
Study objective: This study is planning to develop a new simulation-based ethics education model and evaluate the effectiveness of the model to develop medical students' knowledge, moral reasoning, communication skills, and problem-solving abilities. Several strategies will be conducted to achieve this goal, including faculty development, ethics courses development, and case scenario development.

Methods: The transnational learning and workshops will be arranged for faculty to develop competence for simulation-based ethics education. The workshops will gather the interdisciplinary experts together to discuss and develop the core curriculum and case scenario. The students will be assigned randomly into the simulated clinical ethical situation with simulation patients for the intervention group, and into the workshop discussing clinical ethics case scenario for the control group. The instruments will be developed and the quantitative and qualitative analysis will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* medical students in Kaohsiung Medical University
* agree to participate the study

Exclusion Criteria:

* disagree to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Defining Issues Test (DIT) and self-developed questionnaire | through study completion, an average of 2 years
  Defining Issues Test (DIT) and self-developed questionnaire for evaluation of moral reasoning
ethical decision-making clinical examination | through study completion, an average of 2 years
  clinical scenario exam designed for testing participants' ability of making ethical decision
Problem Identification Test (PIT) and self-developed questionnaire | through study completion, an average of 2 years
  Problem Identification Test (PIT) and self-developed questionnaire for evaluation of moral sensitivity
knowledge test questionnaire | through study completion, an average of 2 years
  questionnaire for ethics knowledge test

SECONDARY OUTCOMES:
results of Objective Structured Clinical Examination | through study completion, an average of 2 years
  test score of Objective Structured Clinical Examination
participant satisfaction questionnaire | through study completion, an average of 2 years
  satisfaction questionnaire for participating the educational activities

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung, Taiwan, Taiwan